CLINICAL TRIAL: NCT01692483
Title: Post-marketing Surveillance Study on the Safety and Effectiveness of Abiraterone Acetate Among Adult Filipino Male Patients With Metastatic Advanced Prostate Cancer
Brief Title: Post-marketing Surveillance Study on the Safety and Effectiveness of Abiraterone Acetate Among Adult Filipino Male Patients With Advanced Metastatic Castration Resistant Prostate Cancer
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor determined study is not required according to PFDA Circular 2013-004
Sponsor: Janssen Pharmaceutica (Industry)
Responsible Party: Sponsor
Other Study IDs: CR100856; 212082PCR4003 (Other: Janssen Pharmaceutica, Philippines)
Record Dates: First submitted 2012-09-21; First posted 2012-09-25 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Prostate Neoplasms
Keywords: Prostate neoplasms; Prostate cancer; Castration resistant prostate cancer; Hormone refractory prostate cancer; Abiraterone acetate; Taxane
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Prednisone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Abiraterone acetate plus prednisone
  Interventions: Drug: Abiraterone acetate; Drug: Prednisone

INTERVENTIONS:
Drug: Abiraterone acetate — Abiraterone 1000 mg (4 x 250 mg tablets) taken orally once daily
Drug: Prednisone — Prednisone or prednisolone 5 mg tablet taken orally twice daily

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of abiraterone acetate in male Filipino patients with advanced metastatic castration resistant prostate cancer (CRPC) who have received prior chemotherapy containing a taxane.

DETAILED DESCRIPTION:
This is an open-label (identity of assigned study drug will be known), observational study to evaluate the safety and efficacy of abiraterone acetate in male Filipino patients with advanced metastatic CRPC who have received prior chemotherapy containing a taxane. Approximately 50 patients will be enrolled. Abiraterone acetate will be administered according to the approved product insert with a low-dose glucocorticoid (prednisone or prednisolone). Patient assessments will be based on the accepted clinical practice in the Philippines. Patients will be monitored for 40 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell histology
* Received at least 1 but not more than 2 cytotoxic chemotherapy regimens for metastatic castration resistant prostate cancer (CRPC) (at least 1 regimen must have contained a taxane such as docetaxel; if a chemotherapy regimen containing a taxane is used more than once, this will be considered as 1 regimen)
* Agrees to protocol-defined use of effective contraception
* Laboratory values within protocol -defined parameters

Exclusion Criteria:

* Serious or uncontrolled co-existent non-malignant disease, including active and uncontrolled infection
* Abnormal liver function
* Uncontrolled hypertension (systolic blood pressure >=160 mmHg or diastolic blood pressure >=95 mmHg)
* Active or symptomatic viral hepatitis or chronic liver disease
* History of pituitary or adrenal dysfunction
* Clinically significant heart disease as evidenced by myocardial infarction, or arterial thrombotic events in the past 6 months, severe or unstable angina, or New York Heart Association (NYHA) Class III or IV heart disease or left ventricular ejection fraction of <50% at baseline
* Known brain metastasis
* History of gastrointestinal disorders (medical disorders or extensive surgery) that may interfere with the absorption of the study drug
* Any acute toxicities due to prior chemotherapy or radiotherapy that have not resolved to a NCI-CTCAE (Version 4.0) Grade of <=1
* Prior systemic treatment with an azole drug (eg, fluconazole, itraconazole, ketoconazole) within 4 weeks of Cycle 1, Day 1
* Condition or situation which, in the investigator's opinion, may put the patient at significant risk, may confound the study results, or may interfere significantly with patient's participation in the study
* Participation in an investigational drug trial within 30 days prior to selection
* Known hypersensitivity to abiraterone acetate, or to any of the components in the formulation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male Filipino patients with advanced metastatic castration resistant prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-07; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants affected by an adverse event | Up to 30 days after the last dose of study medication

SECONDARY OUTCOMES:
Number of patients with disease progression | Baseline up to Week 40

CONTACTS AND LOCATIONS:
Overall Officials: is Janssen Pharmaceutica, Philippines Clinical Trial, Study Director — Janssen Pharmaceutica, Philippines